CLINICAL TRIAL: NCT02421393
Title: Study to Weigh the Effect of Exercise Training on BONE Quality and Strength (SWEET-BONE) in Type 2 Diabetes: an Exercise Intervention Program for Reducing the Risk of Fractures
Brief Title: Study to Weigh the Effect of Exercise Training on BONE (SWEET-BONE) Quality and Strength in Type 2 Diabetes
Acronym: SWEET-BONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Fitness Association, Italy (Other)
Collaborators: University of Roma La Sapienza (Other); S. Andrea Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFA-04
Record Dates: First submitted 2015-04-10; First posted 2015-04-20 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes
Keywords: Bone quality; Bone strength; Fractures; Muscle strength; Gait and balance; Musculo-skeletal symptoms; Falls
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Supervised exercise training on top of standard care (exercise, EXE, group; n=100)
  Interventions: Other: supervised exercise training
- Control (No Intervention): Standard care including advises to maintain a physically active lifestyle, according to current guidelines, by performing any type of commuting, occupational, home and and leisure-time physical activity (PA) (control, CON, group; n=100).

INTERVENTIONS:
Other: supervised exercise training — Two weekly sessions of 75 min each, supervised by an exercise specialist in a dedicated gym facility. Each session will include: 5 min of warm up; 20 min of aerobic training using treadmill; 15 min of resistance training of muscle groups of skeletal sites of fragility fractures; 15 min of "weight bearing" exercises using weighted vests; 8 min of core stability training; 8 min of balance training; and 4 min of flexibility training. Weighted vest worn also during aerobic training and any occupational, home and leisure-time physical activity.
  Arms: Exercise

SUMMARY:
Type 2 diabetes mellitus (T2DM) is associated with increased fracture risk despite normal to increased bone mass, thus suggesting poor bone quality. This study is aimed at weighing the effect of an exercise intervention program on parameters of bone quality in patients with type 2 diabetes mellitus. Two hundred patients with T2DM will be randomized to supervised exercise training on top of standard care (exercise, EXE, group; n=100) versus standard care (control, CON, group; n=100) for 24 months.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is associated with increased fracture risk despite normal to increased bone mass, as assessed as bone mineral density (BMD) by dual-energy X-ray absorptiometry (DXA). Increased fracture risk remains after adjustment for BMD, and also falls, which are more frequent in these individuals than in their non-diabetic counterparts, due to chronic complications and treatments, and for body mass index, which seems to be protective through an increase in BMD. This suggests that patients with T2DM have poor bone quality, i.e. altered bone geometry and microarchitecture, which results in reduced strength. Based on the mechanostat therapy, physical activity (PA)/exercise would be beneficial for preventing fractures in T2DM individuals through greater mechanical loading on the skeleton, which causes favorable bone adaptations, and also by increasing muscle mass, strength, and performance, which reduces the risk of falls by improving gait and balance.

The aim of this study is to assess the effects of a specific exercise training intervention program on parameters of bone quality in patients with type 2 diabetes.

Two hundred patients with T2DM will be randomized to supervised exercise training on top of standard care (exercise, EXE, group; n=100) versus standard care (control, CON, group; n=100) for 24 months.

Sample size calculation is based on a recent report showing that TBS is lower in diabetic vs. control subjects (1.228 vs. 1.298) with a standard deviation of 0.140. To observe a normalization of TBS in EXE participants with a statistical power of 90% (α=0.05) by unpaired t-test, 85 patients per arm are needed (170 total). A sample size of 200 patients will allow to support a dropout rate up to 15%.

A sample of 100 non-diabetic subjects matched 1:2 by age, gender, and BMI will be used as controls for baseline measures.

EXE participants will attend two weekly sessions of 75 min each, supervised by an exercise specialist in a dedicated gym facility. Each session will include: 5 min of warm up; 20 min of aerobic training using treadmill; 15 min of resistance training of muscle groups of skeletal sites of fragility fractures; 15 min of "weight bearing" exercises using weighted vests; 8 min of core stability training; 8 min of balance training; and 4 min of flexibility training. Weighted vest worn also during aerobic training and any occupational, home and leisure-time PA.

CON subjects will receive advises to maintain a physically active lifestyle, according to current guidelines, by performing any type of commuting, occupational, home and leisure-time PA.

All patients will be subjected to a treatment regimen aimed at achieving optimal glycemic, lipid, BP and body weight targets, as established by current guidelines and including glucose-, lipid- and BP-lowering agents as needed. For ethical reasons, drugs will be also adjusted throughout the study to attain target levels and to account for reduced needs. Since all patients are overweight or obese, caloric intake (55% complex carbohydrates, 30% fat, and 15% protein) will be reduced to obtain a negative balance of 500 kcal/day. Requirements will be calculated by adding the estimated energy expenditure from PA to basal metabolism. Adherence to diet will be verified by the use of food diaries and dietary prescriptions will be adjusted at each intermediate visit. Patients with vitamin D levels ranging from 10 to 20 ng/dl will be treated with cholecalciferol 25.000 IU every 2 weeks for 2 months, then with cholecalciferol 25.000 IU every months, whereas those with vitamin D levels ranging from 20 to 30 ng/dl will be given cholecalciferol 25.000 IU every month. At 6 months participants, will be re-evaluated and treatment will be discontinued in case of vitamin D values >30 ng/dl or continued for additional 6 months at the doses indicated above, and so on until the end of the study.

Randomization will be stratified by gender (males versus females), age (65-70 versus 71-75) and type of diabetes treatment (non-insulin versus insulin), using a permuted-block randomization software. Physicians and patients will not be blinded to group assignment, at variance with operators executing instrumental procedures, whereas sample blinding at central laboratory will be achieved using bar codes.

The primary endpoint is the trabecular bone score (TBS), which is derived from the antero-posterior spine raw DXA image(s) from the same region of interest as the BMD measurement by the use of a specific software and correlates with three-dimensional bone micro-architecture parameters. Among the numerous potential measures of bone quality, TBS is the only one that has been consistently shown to be lower in T2DM vs. control subjects.

Secondary endpoints include:

1. other potential measures of bone quality as assessed by peripheral quantitative computed tomography (pQCT) and quantitative ultrasound (QUS);
2. bone mass (BMD as assessed by DXA);
3. bone metabolism (sclerostin and other biochemical markers of bone formation and resorption);
4. body composition (total body lean and fat mass by total body DXA);
5. muscle strength (by dynamometer);
6. muscle mass/density (by pQCT);
7. balance, gait and power (by Short Battery Performance Test);
8. musculoskeletal (MS) symptoms (by questionnaire);

h. number of falls (by questionnaire); i. symptomatic and asymptomatic fractures (by history or medical records and vertebral morphometry, respectively).

Other measures include:

* quality of life (QoL);
* cardiorespiratory fitness;
* flexibility;
* volume of PA;
* coronary heart disease 10-year risk score.

Dietary intake and adverse events will be also recorded. Participants from both groups will be followed for additional 5 years in order to record the number of falls and eventual fractures during this time period. PA and MS symptoms will be also monitored throughout this 5-year interval. To this end, patients will be seen yearly (or every 6 months according to the degree of glycemic control and the overall cardiovascular risk profile) in order to collect self-report data on number of falls and type and amount of PA from a daily diary, clinical documentation on eventual fractures, and MS questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* diabetes duration >5-year
* sedentary lifestyle (i.e. more than 8 hours/day spent in any waking behavior characterized by an energy expenditure ≤1.5 metabolic equivalents [METs] while in a sitting or reclining posture) from at least 6 months;
* physically inactivity (i.e. insufficient amounts of physical activity [PA] according to current guidelines) from at least 6 months;
* body mass index (BMI) 27-40 kg/m2;
* ability to walk 1.6 Km without assistance;
* a Short Battery Performance Test score ranging from 4 to 9;
* eligibility after cardiologic evaluation.

Exclusion Criteria:

* any condition limiting participation in a clinical trial, including psychiatric disorders or hospitalization for depression in the past 6 months;
* any condition limiting PA/exercise, including musculoskeletal disorders or deformities, central nervous system dysfunction such as hemiparesis, myelopathies, cerebral ataxia, vestibular dysfunction, and postural hypotension (i.e. a fall of >20 mmHg of systolic or >10 mmHg of diastolic blood pressure when changing position);
* cancer and other life-expectancy limiting conditions;
* recent major acute cardiovascular event, including heart attack, stroke/transient ischemic attack(s), revascularization procedure, or participation in a cardiac rehabilitation program within the past three months, or documented history of pulmonary embolism in the past six months;
* pre-proliferative and proliferative retinopathy;
* macroalbuminuria and/or estimated glomerular filtration rate (eGFR) <45 ml/min/1.73 m2;
* ankle/brachial index (ABI) <0.9;
* severe motor and sensory neuropathy;
* diabetic foot with history of ulcer;
* hemoglobin (Hb) A1c >9.0%;
* blood pressure (BP) >150/90 mmHg;
* vitamin D <10 ng/ml;
* treatment with anti-fracturative agents, estrogens, aromatase inhibitors, testosterone, corticosteroids and/or glitazon;
* previous documented non-traumatic fractures,
* total spine deformity index (SDI) >3 (and >1 in a single vertebra);
* a T score <-2.5 at spine/hip at dual-energy X-ray absorptiometry (DXA). Subjects with HbA1c or blood pressure above the indicated threshold will be receive appropriate treatment and will be re-evaluated after 3 months. Patients with vitamin D levels < 10 ng/dl will be treated with cholecalciferol 25.000 IU/week for 6 weeks and will be re-evaluated for eligibility 2 weeks after the last

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Effect of intervention on bone quality (trabecular bone score) | 2 years
  Effect of exercise intervention training on trabecular bone score (TBS)

SECONDARY OUTCOMES:
Effect of intervention on other measures of bone quality (composite) | 2 years
  Effect of exercise intervention training on peripheral quantitative computed tomography (pQCT) and quantitative ultrasound (QUS) parameters
Effect of intervention on bone mass (dual-energy X-ray absorptiometry) | 2 years
  Effect of exercise intervention training on bone mineral density (BMD) as assessed by dual-energy X-ray absorptiometry (DXA)
Effect of intervention on bone metabolism (composite) | 2 years
  Effect of exercise intervention training on biochemical markers of bone formation and resorption
Effect of intervention on body composition (total body dual-energy X-ray absorptiometry ) | 2 years
  Effect of exercise intervention training on total body lean and fat mass as assessed by total body dual-energy X-ray absorptiometry (DXA)
Effect of intervention on muscle strength (dynamometry) | 2 years
  Effect of exercise intervention training on muscle strength as assessed by dynamometer
Effect of intervention on muscle mass/density (pQcT) | 2 years
  Effect of exercise intervention training on muscle mass/density as assessed by pQCT
Effect of intervention on balance, gait and power (Short Battery Performance Test) | 2 years
  Effect of exercise intervention training on a composite score of for balance, gait and power as assessed by Short Battery Performance Test
Effect of intervention on on musculoskeletal (MS) symptoms (questionnaire) | 7 years
  Effect of exercise intervention training oon musculoskeletal (MS) symptoms as assessed by the use of a questionnaire
Effect of intervention on number of falls (self-report daily diary) | 7 years
  Effect of exercise intervention training on number of falls as assessed by the use of a self-report daily diary
Effect of intervention on fracture incidence (history or medical records and vertebral morphometry) | 2-7 years
  Effect of exercise intervention training on the incidence of symptomatic and asymptomatic fractures as assessed by history or medical records and vertebral morphometry, respectively

OTHER OUTCOMES:
Effect of intervention on quality of life (QoL) (SF-36 questionnaire) | 2 years
  Effect of exercise intervention training on quality of life (QoL) as assessed by SF-36 questionnaire
Effect of intervention on cardiorespiratory fitness (VO2max) | 2 years
  Effect of exercise intervention training on cardiorespiratory fitness as assessed by maximal oxygen consumption (VO2max)
Effect of intervention on flexibility (bending test) | 2 years
  Effect of exercise intervention training on hip and trunk flexibility as assessed by bending test
Effect of intervention on volume of physical activity (PA) (self-report daily diary) | 7 years
  Effect of exercise intervention training on volume of physical activity (PA) as assessed by self-report daily diary
Effect of intervention on coronary heart disease 10-year risk | 2 years
  Effect of exercise intervention training on cardiovascular risk profile as assessed by on coronary heart disease 10-year risk calculated from clinical and biochemical measurements

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pugliese, MD, PhD, Principal Investigator — University of Roma La Sapienza; Francesco Conti, MD, PhD, Study Director — University of Roma La Sapienza
Locations (1):
- S. Andrea Hospital, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balducci S, Zanuso S, Cardelli P, Salvi L, Mazzitelli G, Bazuro A, Iacobini C, Nicolucci A, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Changes in physical fitness predict improvements in modifiable cardiovascular risk factors independently of body weight loss in subjects with type 2 diabetes participating in the Italian Diabetes and Exercise Study (IDES). Diabetes Care. 2012 Jun;35(6):1347-54. doi: 10.2337/dc11-1859. Epub 2012 Mar 7. PMID 22399699
- [Background] Balducci S, Zanuso S, Nicolucci A, De Feo P, Cavallo S, Cardelli P, Fallucca S, Alessi E, Fallucca F, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Effect of an intensive exercise intervention strategy on modifiable cardiovascular risk factors in subjects with type 2 diabetes mellitus: a randomized controlled trial: the Italian Diabetes and Exercise Study (IDES). Arch Intern Med. 2010 Nov 8;170(20):1794-803. doi: 10.1001/archinternmed.2010.380. PMID 21059972
- [Background] Bonds DE, Larson JC, Schwartz AV, Strotmeyer ES, Robbins J, Rodriguez BL, Johnson KC, Margolis KL. Risk of fracture in women with type 2 diabetes: the Women's Health Initiative Observational Study. J Clin Endocrinol Metab. 2006 Sep;91(9):3404-10. doi: 10.1210/jc.2006-0614. Epub 2006 Jun 27. PMID 16804043
- [Background] Burghardt AJ, Issever AS, Schwartz AV, Davis KA, Masharani U, Majumdar S, Link TM. High-resolution peripheral quantitative computed tomographic imaging of cortical and trabecular bone microarchitecture in patients with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2010 Nov;95(11):5045-55. doi: 10.1210/jc.2010-0226. Epub 2010 Aug 18. PMID 20719835
- [Background] Carnevale V, Romagnoli E, D'Erasmo L, D'Erasmo E. Bone damage in type 2 diabetes mellitus. Nutr Metab Cardiovasc Dis. 2014 Nov;24(11):1151-7. doi: 10.1016/j.numecd.2014.06.013. Epub 2014 Jul 27. PMID 25150773
- [Background] Chan MY, Frost SA, Center JR, Eisman JA, Nguyen TV. Relationship between body mass index and fracture risk is mediated by bone mineral density. J Bone Miner Res. 2014 Nov;29(11):2327-35. doi: 10.1002/jbmr.2288. PMID 24862213
- [Background] Cousins JM, Petit MA, Paudel ML, Taylor BC, Hughes JM, Cauley JA, Zmuda JM, Cawthon PM, Ensrud KE; Osteoporotic Fractures in Men (MrOS) Study Group. Muscle power and physical activity are associated with bone strength in older men: The osteoporotic fractures in men study. Bone. 2010 Aug;47(2):205-11. doi: 10.1016/j.bone.2010.05.003. Epub 2010 May 11. PMID 20466088
- [Background] De Laet C, Kanis JA, Oden A, Johanson H, Johnell O, Delmas P, Eisman JA, Kroger H, Fujiwara S, Garnero P, McCloskey EV, Mellstrom D, Melton LJ 3rd, Meunier PJ, Pols HA, Reeve J, Silman A, Tenenhouse A. Body mass index as a predictor of fracture risk: a meta-analysis. Osteoporos Int. 2005 Nov;16(11):1330-8. doi: 10.1007/s00198-005-1863-y. Epub 2005 Jun 1. PMID 15928804
- [Background] de Waard EA, van Geel TA, Savelberg HH, Koster A, Geusens PP, van den Bergh JP. Increased fracture risk in patients with type 2 diabetes mellitus: an overview of the underlying mechanisms and the usefulness of imaging modalities and fracture risk assessment tools. Maturitas. 2014 Nov;79(3):265-74. doi: 10.1016/j.maturitas.2014.08.003. Epub 2014 Aug 18. PMID 25192916
- [Background] Dobnig H, Piswanger-Solkner JC, Roth M, Obermayer-Pietsch B, Tiran A, Strele A, Maier E, Maritschnegg P, Sieberer C, Fahrleitner-Pammer A. Type 2 diabetes mellitus in nursing home patients: effects on bone turnover, bone mass, and fracture risk. J Clin Endocrinol Metab. 2006 Sep;91(9):3355-63. doi: 10.1210/jc.2006-0460. Epub 2006 May 30. PMID 16735485
- [Background] Donnelly E. Methods for assessing bone quality: a review. Clin Orthop Relat Res. 2011 Aug;469(8):2128-38. doi: 10.1007/s11999-010-1702-0. PMID 21116752
- [Background] Gonnelli S, Caffarelli C, Nuti R. Obesity and fracture risk. Clin Cases Miner Bone Metab. 2014 Jan;11(1):9-14. doi: 10.11138/ccmbm/2014.11.1.009. PMID 25002873
- [Background] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Background] Janghorbani M, Van Dam RM, Willett WC, Hu FB. Systematic review of type 1 and type 2 diabetes mellitus and risk of fracture. Am J Epidemiol. 2007 Sep 1;166(5):495-505. doi: 10.1093/aje/kwm106. Epub 2007 Jun 16. PMID 17575306
- [Background] Johansson H, Kanis JA, Oden A, McCloskey E, Chapurlat RD, Christiansen C, Cummings SR, Diez-Perez A, Eisman JA, Fujiwara S, Gluer CC, Goltzman D, Hans D, Khaw KT, Krieg MA, Kroger H, LaCroix AZ, Lau E, Leslie WD, Mellstrom D, Melton LJ 3rd, O'Neill TW, Pasco JA, Prior JC, Reid DM, Rivadeneira F, van Staa T, Yoshimura N, Zillikens MC. A meta-analysis of the association of fracture risk and body mass index in women. J Bone Miner Res. 2014 Jan;29(1):223-33. doi: 10.1002/jbmr.2017. PMID 23775829
- [Background] Kim JH, Choi HJ, Ku EJ, Kim KM, Kim SW, Cho NH, Shin CS. Trabecular bone score as an indicator for skeletal deterioration in diabetes. J Clin Endocrinol Metab. 2015 Feb;100(2):475-82. doi: 10.1210/jc.2014-2047. Epub 2014 Nov 4. PMID 25368976
- [Background] Leslie WD, Aubry-Rozier B, Lamy O, Hans D; Manitoba Bone Density Program. TBS (trabecular bone score) and diabetes-related fracture risk. J Clin Endocrinol Metab. 2013 Feb;98(2):602-9. doi: 10.1210/jc.2012-3118. Epub 2013 Jan 22. PMID 23341489
- [Background] Leslie WD, Rubin MR, Schwartz AV, Kanis JA. Type 2 diabetes and bone. J Bone Miner Res. 2012 Nov;27(11):2231-7. doi: 10.1002/jbmr.1759. Epub 2012 Sep 28. PMID 23023946
- [Background] Martyn-St James M, Carroll S. Effects of different impact exercise modalities on bone mineral density in premenopausal women: a meta-analysis. J Bone Miner Metab. 2010 May;28(3):251-67. doi: 10.1007/s00774-009-0139-6. Epub 2009 Dec 15. PMID 20013013
- [Background] Napoli N, Strotmeyer ES, Ensrud KE, Sellmeyer DE, Bauer DC, Hoffman AR, Dam TT, Barrett-Connor E, Palermo L, Orwoll ES, Cummings SR, Black DM, Schwartz AV. Fracture risk in diabetic elderly men: the MrOS study. Diabetologia. 2014 Oct;57(10):2057-65. doi: 10.1007/s00125-014-3289-6. Epub 2014 Jun 9. PMID 24908567
- [Background] Park SW, Goodpaster BH, Strotmeyer ES, de Rekeneire N, Harris TB, Schwartz AV, Tylavsky FA, Newman AB. Decreased muscle strength and quality in older adults with type 2 diabetes: the health, aging, and body composition study. Diabetes. 2006 Jun;55(6):1813-8. doi: 10.2337/db05-1183. PMID 16731847
- [Background] Petit MA, Paudel ML, Taylor BC, Hughes JM, Strotmeyer ES, Schwartz AV, Cauley JA, Zmuda JM, Hoffman AR, Ensrud KE; Osteoporotic Fractures in Men (MrOs) Study Group. Bone mass and strength in older men with type 2 diabetes: the Osteoporotic Fractures in Men Study. J Bone Miner Res. 2010 Feb;25(2):285-91. doi: 10.1359/jbmr.090725. PMID 19594301
- [Background] Schwartz AV, Hillier TA, Sellmeyer DE, Resnick HE, Gregg E, Ensrud KE, Schreiner PJ, Margolis KL, Cauley JA, Nevitt MC, Black DM, Cummings SR. Older women with diabetes have a higher risk of falls: a prospective study. Diabetes Care. 2002 Oct;25(10):1749-54. doi: 10.2337/diacare.25.10.1749. PMID 12351472
- [Background] Schwartz AV, Sellmeyer DE, Ensrud KE, Cauley JA, Tabor HK, Schreiner PJ, Jamal SA, Black DM, Cummings SR; Study of Osteoporotic Features Research Group. Older women with diabetes have an increased risk of fracture: a prospective study. J Clin Endocrinol Metab. 2001 Jan;86(1):32-8. doi: 10.1210/jcem.86.1.7139. PMID 11231974
- [Background] Tao B, Liu JM, Zhao HY, Sun LH, Wang WQ, Li XY, Ning G. Differences between measurements of bone mineral densities by quantitative ultrasound and dual-energy X-ray absorptiometry in type 2 diabetic postmenopausal women. J Clin Endocrinol Metab. 2008 May;93(5):1670-5. doi: 10.1210/jc.2007-1760. Epub 2008 Mar 4. PMID 18319321
- [Background] Vestergaard P. Discrepancies in bone mineral density and fracture risk in patients with type 1 and type 2 diabetes--a meta-analysis. Osteoporos Int. 2007 Apr;18(4):427-44. doi: 10.1007/s00198-006-0253-4. Epub 2006 Oct 27. PMID 17068657
- [Derived] Balducci S, Conti F, Sacchetti M, Russo CR, Argento G, Haxhi J, Orlando G, Rapisarda G, D'Errico V, Cardelli P, Pugliese L, Laghi A, Vitale M, Bollanti L, Zanuso S, Nicolucci A, Pugliese G; SWEET BONE Investigators. Study to Weigh the Effect of Exercise Training on BONE quality and strength (SWEET BONE) in type 2 diabetes: study protocol for a randomised clinical trial. BMJ Open. 2019 Nov 4;9(11):e027429. doi: 10.1136/bmjopen-2018-027429. PMID 31690602
- See also: Web site of the Metabolic Fitness Association — http://www.metabolicfitness.it/